CLINICAL TRIAL: NCT07264088
Title: The FOLLOW UP Study - a Natural Experiment Estimating the Clinical and Cost-effectiveness of Follow up Strategies After Curative Treatment for Prostate Cancer
Brief Title: Identifying the Best Follow up Approach for People Who Have Had Treatment to Cure Newly Diagnosed Prostate Cancer
Acronym: FOLLOW-UP
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University of Aberdeen (Other); University of Leeds (Other); Cardiff University (Other); University of Sheffield (Other); University of Southampton (Other); University College, London (Other); Royal Marsden NHS Foundation Trust (Other); North Bristol NHS Trust (Other); Cardiff and Vale University Health Board (Other Government); Liverpool University Hospitals NHS Foundation Trust (Other Government); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 181848; NIHR150376 (Other Grant/Funding Number: NIHR HTA); 342362 (Other: IRAS); 25/LO/0753 (Other: London - Chelsea Research Ethics Committee); 25_CAG_0127 (Other: Confidentiality Advisory Group)
Record Dates: First submitted 2025-09-30; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate cancer after curative treatment; prostate cancer follow up; propensity-matched cohort study; qualitative; discrete choice experiment; economic evaluation; routine data; patient survey
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Self-Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hospital based follow up: Exclusively hospital led follow up, face-to-face or remotely by the specialist treating team.
  Interventions: Other: Hospital based follow up
- Primary care based follow up: After the initial hospital follow up, patients are discharged and exclusively managed by (non-specialist) general practices (GP or nurse led) in face-to-face or remote appointments, with hospital referral as necessary.
  Interventions: Other: Primary care based follow up
- Planned shared care follow up: An ongoing combination of general practice and hospital management
  Interventions: Other: Planned shared care follow up
- Self-management: After initial hospital follow up, patients are discharged and managed remotely, with no scheduled review. A tracking system monitors prostate-specific antigen (PSA) tests performed in primary care or secondary care. Patients access support workers for remote consultation to discuss symptoms and request further specialist management as required.
  Interventions: Other: Self-management

INTERVENTIONS:
Other: Hospital based follow up — Exclusively hospital led follow up, face-to-face or remotely by the specialist treating team.
  Groups: Hospital based follow up
Other: Primary care based follow up — After the initial hospital follow up, patients are discharged and exclusively managed by (non-specialist) general practices (GP or nurse led) in face-to-face or remote appointments, with hospital referral as necessary.
  Groups: Primary care based follow up
Other: Planned shared care follow up — An ongoing combination of general practice and hospital management
  Groups: Planned shared care follow up
Other: Self-management — After initial hospital follow up, patients are discharged and managed remotely, with no scheduled review. A tracking system monitors prostate-specific antigen (PSA) tests performed in primary care or secondary care. Patients access support workers for remote consultation to discuss symptoms and request further specialist management as required.
  Groups: Self-management

SUMMARY:
Over 20,000 patients a year in the UK get surgery or radiotherapy to cure their prostate cancer. These men then undergo regular check-ups to manage potential side effects and see if cancer recurs so it can be treated quickly. The organisation of these check-ups varies across the country as it is not known which approach is best. The four different established approaches are (i) check-ups performed in hospital outpatients by the same team that provided treatment; (ii) patients seen regularly by their GP with hospital referral as necessary; (iii) planned shared care between general practice and hospital follow up; or (iv) patients supported to provide checks on themselves (self-care) and reaching out to a doctor or a nurse when required. This study will compare these options to establish which is best for patients and makes the best use of the NHS resources.

DETAILED DESCRIPTION:
This is a pragmatic, prospective, propensity-matched, cohort study using routine data, with an embedded patient survey, economic evaluation, and qualitative and preference studies. Individual sites will be classified according to one of the four follow up strategies to compare outcomes in a natural experiment. Individual participants will be clustered within their treating hospital.

The main cohort for the study will be identified from the National Disease Registration Service Cancer Registry. Data on treatments, diagnoses, clinic attendances and other events that occur in secondary care from 3 years prior to diagnosis will be extracted from databases linked to the Cancer Registry including Cancer Pathway, Radiotherapy Dataset (RTDS), Systemic Anti-Cancer dataset (SACT) and Hospital Episode Statistics (HES). These datasets are referred to collectively as 'HES-linked data'. HES-linked data will be collected from 3 years prior to diagnosis, to enable analyses to be adjusted for patient medical history and pattern of health service use prior to diagnosis with prostate cancer, to the latest available date (expected to be 31 December 2026).

To identify the most clinically and cost-effective follow up strategy for patients, five interrelated work packages (WPs) will address specific objectives:

- WP1: Determine safety and clinical effectiveness of different follow up strategies

Stage 1: The utility of HES-linked data to study treatment for prostate cancer recurrence will be validated. It will be confirmed if databases contain the parameters required and are complete enough to robustly assess outcomes in secondary care including time to treatment for cancer recurrence and treatment for side-effects from primary treatment. Detailed statistical methods and computer code will be developed for determining whether follow up strategies are equivalent for treatment of recurrence, including methods for dealing with missing patients and treatment variables. A preliminary investigation of hospital adherence to stated follow up strategies will be conducted.

Stage 2: All primary and secondary outcomes will be measured using both HES-linked datasets and information collected through the patient survey in WP2. The methods developed in stage 1 will be used to assess the equivalence of the four follow up strategies for the primary outcome of treatment for cancer recurrence at 3 years, the key secondary outcome of time to hospital treatment for cancer recurrence, and remaining secondary outcomes.

-WP2: Measure side effects of prostate cancer treatments, patient quality of life and recurrence outcomes not captured in routine data

A survey will be designed and administered to capture data from a subgroup of study participants on adverse effects of initial cancer treatment, how those adverse effects were managed, health service utilisation and HRQoL. The survey will ask patients whether and when they received hormone therapy for prostate cancer recurrence, providing data for WP1 on recurrence treatments not captured in HES-linked databases.

-WP3: Identify key patient perspectives on the important features of follow-up

A qualitative interview study will be conducted with patients with lived experience of prostate cancer and follow up, purposively sampling geographic spread, socioeconomic class and ethnicity (WP3 is sponsored by University of Aberdeen and is described in a separate protocol and has separate ethics approvals). Early findings will inform the design of the Discrete Choice Experiment (DCE) to be deployed in WP5.

-WP4: Evaluate the cost-effectiveness of each follow up strategy

The use of primary and secondary health care services during follow up to estimate the costs of the four follow up strategies will be assessed using HES-linked and patient survey data. An economic evaluation model will be developed to compare the patient lifetime costs and outcomes of the four strategies, and identify the approach that provides the best value for money for the NHS.

-WP5: Define patient preferences for follow-up

A DCE will be conducted to understand how patients might respond to follow up strategies with different attributes and elicit patient preferences. Questions for the DCE will be designed using early qualitative findings (WP3) and will be included as a module in the patient survey (WP2) for a subgroup of survey recipients.

ELIGIBILITY:
Inclusion criteria:

All hospitals in England that provide radical prostatectomy or radical radiotherapy or focal therapy for prostate cancer and are identified by clinicians as receiving one of the four follow up strategies of interest will be eligible for inclusion in the study.

Individual patients satisfying the following criteria will be eligible for inclusion:

* Having newly-diagnosed non-metastatic, clinically localised prostate cancer (ICD-10 code C61) in the Cancer Registry between 1 January 2018 and 31 December 2023;
* Age 18 or over at diagnosis;
* Completed primary curative treatment at an eligible hospital between 1 January 2019 and 31 December 2023 with either: radical radiotherapy +/- hormones, or radical prostatectomy with curative intent +/- lymphadenectomy, or focal therapy, in keeping with local practice;
* Alive with no disease progression or metastasis 6 months after the date of completion of primary curative treatment.

Exclusion criteria:

* Men who are treated for metastatic cancer; or receiving palliative prostate cancer care;
* Men who have opted out of their data being used as part of national routine data sets will be excluded (https://digital.nhs.uk/services/national-data-opt-out).

Recruitment to the survey component of the study will be limited to a sub-cohort of eligible participants that additionally meet the following criteria:

* Alive;
* Have achieved between three to four and a half years of follow up (from completion of initial curative treatment) during the survey period.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men aged 18 and over who were newly diagnosed with prostate cancer between January 2018 and December 2023 and completed curative treatment to cure their prostate cancer at a hospital in England between January 2019 and December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Safety and clinical effectiveness defined by treatment for cancer recurrence | At 3 years following end of initial radical surgery or radiotherapy or focal therapy
  Probability of cancer recurrence treatment calculated from analysis of time to recurrence treatment, measured using Hospital Episode Statistics (HES)-linked cancer databases and patient survey that includes domains on cancer recurrence and treatment.
Estimate cost-effectiveness | At 3 years, extrapolated over the remaining patient lifetime
  Modelled cost-effectiveness reported as incremental cost per quality adjusted life year (QALY) gained at different points over patient lifetime from an NHS and personal social services perspective, measured using HES-linked databases and patient survey

SECONDARY OUTCOMES:
Time to treatment for cancer recurrence provided in secondary care | Up to 7 complete years following end of initial radical surgery or radiotherapy or focal therapy
  Restricted mean time to treatment for cancer recurrence provided in secondary care, measured using HES-linked databases.
Metastases, cancer specific and overall survival | Up to 7 complete years following end of initial radical surgery or radiotherapy or focal therapy
  Time to metastasis, time to prostate cancer specific death, and overall survival (including time to and cause of non-prostate cancer deaths), measured using HES-linked databases
Cancer recurrence treatments (salvage to cure vs palliative suggesting delayed diagnosis) | Up to 3 years following end of initial radical surgery or radiotherapy or focal therapy
  A binary outcome (cancer recurrence treatment) that takes the value 1 if the recurrence treatment was salvage with intent to cure and 0 if the recurrence treatment was palliative. This will be assessed using the type of first treatment received for recurrence, as recorded in HES-linked databases or reported in the patient survey.
Health related quality of life (HRQoL) | At 3 to 4.5 years following end of initial radical surgery or radiotherapy or focal therapy
  The EuroQol 5-Dimension 5-Level (EQ-5D-5L) instrument will be used to measure HRQoL in the patient survey. The EQ-5D-5L index values range from a minimum of -0.594 (representing health states considered worse than death) to a maximum of 1.000 (representing full health). In this scoring system, higher values indicate better health-related quality of life outcomes.
Health related quality of life (HRQoL) | At 3 to 4.5 years following end of initial radical surgery or radiotherapy or focal therapy
  The Expanded Prostate Cancer Index Composite 26-item short form (EPIC-26) is collected in the patient survey and measures prostate cancer-specific HRQoL across four domains: urinary, bowel, sexual and hormonal function. Scores for each domain are transformed to a 0-100 scale, where higher values indicate better HRQoL (reflecting less symptom burden and greater functional well-being).
Physical and psychological complications of treatment | At 3 years following end of initial radical surgery or radiotherapy or focal therapy
  Including those resulting in specialist referrals or prescribing, measured using HES-linked databases and patient survey
Prostate cancer core outcome set (COS) | At 3 years following end of initial radical surgery or radiotherapy or focal therapy
  COS measures relevant to follow up and treatment not otherwise captured: perioperative deaths, positive surgical margin, thromboembolic disease, urethral stricture and side-effects of hormonal therapy, measured using patient survey and HES-linked databases.
Patient experience and satisfaction | For the qualitative study: At enrolment for the qualitative study. For the DCE: At 3 to 4.5 years following end of initial radical surgery or radiotherapy or focal therapy
  Measured from the Discrete Choice Experiment (DCE). DCE reported as % uptake of follow-up with minimum score 0% and maximum score 100%.
Adherence to follow up strategy | At 3 years following end of initial radical surgery or radiotherapy or focal therapy
  Level of adherence to each follow up strategy is based on outpatient clinic attendance recorded in HES-linked databases and GP attendance reported in the patient survey. Measurement will involve counts of appointments from both sources combined and compared with the expected count based on the follow up strategy in use at each participating centre. For each treatment type (surgery, radiotherapy and focal therapy) a measure of adherence will be derived and reported. Full details will be developed and reported in the Statistical Analysis Plan before data analysis.
Costs to health services | Measured at up to 7 years as well as at 3 years (for consistency with the key primary and secondary outcomes estimated in work package 1), following end of initial radical surgery or radiotherapy or focal therapy.
  Total cost of health services used in primary and secondary care, measured using HES-linked databases and patient survey.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Heer, BMed Sci MB BS MRCS PhD FRCS, Principal Investigator — Imperial College London
Locations (1):
- London School of Hygiene & Tropical Medicine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
In development